CLINICAL TRIAL: NCT01284816
Title: Impact of Bariatric Surgery on Epicardial Adipose Tissue and on Myocardial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: None
Other Study IDs: 2010-A00696-33
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Severely Obese Patients
Keywords: severely obese patients
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- severely obese patients (Other): 35 patients addressed for severe obesity in the Endocrinology department of Marseille North Hospital before (V1) and 6 months (V2) after bariatric surgery
  Interventions: Procedure: bariatric surgery

INTERVENTIONS:
Procedure: bariatric surgery — The bariatric surgery is a relevant treatment for severely obese patients those with metabolic complications, as it significantly reduces weight, hypertension and ameliorates glycemic control.

SUMMARY:
Growing evidence suggests that bariatric surgery is a relevant treatment for severely obese patients, especially those with metabolic complications, as it significantly reduces weight, hypertension and ameliorates glycemic control. Its action on adipose tissue distribution and in particular on epicardial adipose tissue EAT remains unknown. Whether metabolic improvement is associated with EAT reduction is also unknown.

The researchers thus investigated the effect of bariatric surgery on EAT in severely obese patients. The primary endpoint of this study was the change in EAT amount 6 months after bariatric surgery.

DETAILED DESCRIPTION:
The best of our knowledge, no study has really addressed whether this EAT was modulated by diet or therapeutics like bariatric surgery. The researchers were particularly interested in studying the impact of bariatric surgery and of weight loss on the amount of EAT and whether reduction in EAT could have a positive impact on myocardial function.

ELIGIBILITY:
Inclusion Criteria:

* men or women who have more than 18 years
* patients have been informed and have consented
* severely obese patients with surgery indication

Exclusion Criteria:

* contraindications at surgery, at MNR imagery
* History of infarct, of congenital cardiomyopathy
* Treatment modifying the distribution of the fat
* Pregnant or breast-feeding women
* patients less than 18 years
* Patient without consentment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-09; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The change in EAT amount 6 months after bariatric surgery. | 36 months
  We thus investigated the effect of bariatric surgery on EAT in severely obese patients.

SECONDARY OUTCOMES:
Evaluation of 3 parameters | 36 months
  1. to evaluate the variation in myocardial, hepatic , pancreatic and triglyceride content
  2. to evaluate the variation in left ventricular function or myocardial function
  3. and to describe the relationships between changes in visceral abdominal fat, subcutaneous fat and epicardial fat

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dutour, Professor, Principal Investigator — AP-HM
Locations (1):
- AP-HM, Marseille, France

REFERENCES:
- [Derived] Soghomonian A, Dutour A, Kachenoura N, Thuny F, Lasbleiz A, Ancel P, Cristofari R, Jouve E, Simeoni U, Kober F, Bernard M, Gaborit B. Is increased myocardial triglyceride content associated with early changes in left ventricular function? A 1H-MRS and MRI strain study. Front Endocrinol (Lausanne). 2023 Jun 22;14:1181452. doi: 10.3389/fendo.2023.1181452. eCollection 2023. PMID 37424866
- [Derived] Henry JA, Abdesselam I, Deal O, Lewis AJ, Rayner J, Bernard M, Dutour A, Gaborit B, Kober F, Soghomonian A, Sgromo B, Byrne J, Bege T, Neubauer S, Borlaug BA, Rider OJ. Changes in epicardial and visceral adipose tissue depots following bariatric surgery and their effect on cardiac geometry. Front Endocrinol (Lausanne). 2023 Jan 25;14:1092777. doi: 10.3389/fendo.2023.1092777. eCollection 2023. PMID 36761185
- [Derived] Gaborit B, Jacquier A, Kober F, Abdesselam I, Cuisset T, Boullu-Ciocca S, Emungania O, Alessi MC, Clement K, Bernard M, Dutour A. Effects of bariatric surgery on cardiac ectopic fat: lesser decrease in epicardial fat compared to visceral fat loss and no change in myocardial triglyceride content. J Am Coll Cardiol. 2012 Oct 9;60(15):1381-9. doi: 10.1016/j.jacc.2012.06.016. Epub 2012 Aug 29. PMID 22939560